CLINICAL TRIAL: NCT05134909
Title: Custom Vision-Corrective Lens Study
Brief Title: Customized Contact Lenses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Geunyoung Yoon, Professor, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00003195
Record Dates: First submitted 2021-11-11; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study: Keratoconus (Experimental): Customized contact lenses will be fitted to each study subject based on their own optical defects.
  Interventions: Device: Customized contact lens

INTERVENTIONS:
Device: Customized contact lens — The customized lenses are designed to correct the eye's optical aberrations.

SUMMARY:
The overall goal of this project is to improve the visual quality of individuals who have abnormal corneal conditions that alter the shape of their cornea (eg. keratoconus). Patients with an abnormal corneal shape have substantial lower and higher order aberrations (distortions in the eye). This results in reduced visual acuity which cannot be corrected by regular sphero-cylindrical correction. Compensating for these aberrations has been challenging due to difficulty measuring their wavefront aberrations accurately and, consequently, manufacturing the custom contact lenses with irregular optical profiles. This project is designed to systematically overcome these obstacles with a customized scleral and/or soft contact lens capable of compensating for the lower and higher order aberrations of the eye.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and understand the informed consent document in English
* 18 to 75 years of age
* Received diagnosis of keratoconus by a clinician
* Willing and able to follow instructions

Exclusion Criteria:

* Has best corrected visual acuity of 20/20 or better in the keratoconic eye(s).
* Normal/typical subjects
* Is unable to handle, insert, remove or care for the study lenses.
* Has any active anterior segment disease, pathology, or surgery affecting vision, refraction, or the ability to wear a contact lens
* History of ocular pharmacological treatment
* History of ocular trauma or surgery causing abnormal corneal curvature or distorted vision History of contact lens intolerance
* Pregnant at the time of enrollment in the study (self-reported- It has been shown hormonal changes during pregnancy may affect corneal biomechanics negatively)
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers under the age of 18 because it has been shown the average age of the appearance of Keratoconus is the second decade of life ( 15-18 years of age)
* Prisoners

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | up to 2 months
  Snellen "Tumbling E" method will be used to determine the smallest visible letter that a subject can see.
Contrast sensitivity | up to 2 months
  Light and dark sinusoidal stripes (Gabor gratings) will used to determine the smallest contrast that a subject can see.

CONTACTS AND LOCATIONS:
Overall Officials: Geunyoung Yoon, PhD, Principal Investigator — University of Houston

IPD SHARING:
Plan to Share IPD: No